CLINICAL TRIAL: NCT00975793
Title: A Multi-centre, Randomised Controlled Trial of Early Goal-directed Therapy in Patients Presenting to the Emergency Department With Severe Sepsis in Australasia
Brief Title: Australasian Resuscitation In Sepsis Evaluation Randomised Controlled Trial
Acronym: ARISE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belinda Howe (Other)
Collaborators: Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); Australasian College for Emergency Medicine (Other)
Responsible Party: Sponsor-Investigator, Belinda Howe, Project manager, ANZIC- Research Centre, Monash University, Monash University
Organization: Monash University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZIC - RC/RB001; NHMRC Project grant no. 491075
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Severe Sepsis
Keywords: Sepsis; Severe sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Randomised allocation of standard care at the clinician's discretion in accordance with current best practice.
- Early Goal Directed Therapy (Experimental): Randomised allocation of early goal-directed therapy (EGDT).
  Interventions: Other: Early Goal Directed Therapy (EGDT)

INTERVENTIONS:
Other: Early Goal Directed Therapy (EGDT) — Randomised allocation of early goal-directed therapy (EGDT). EGDT involves treatment with intravenous fluids, and medications to support the blood pressure and heart following a protocol. A special catheter is inserted to monitor central blood oxygen levels and the standard treatments are given according to the blood oxygen level reading. EGDT is given for 6 hours, then the patient receives standard care.
  Arms: Early Goal Directed Therapy

SUMMARY:
The ARISE RCT is a multi-centre, randomised, controlled trial of EGDT compared to standard care in patients with severe sepsis presenting to the ED. The study will be conducted in multiple sites with 1600 patients enrolled into the study.

Hypothesis to be tested: EGDT, compared to standard Australasian resuscitation practice, reduces 90-day all-cause mortality in patients presenting to the ED with severe sepsis.

DETAILED DESCRIPTION:
The primary aim of the study is to determine whether providing EGDT, compared to standard care, reduces 90-day mortality in patients presenting to the ED of hospitals in Australasia with severe sepsis.

Each patient meeting all of the exclusion criteria and none of the exclusion criteria will be randomised in the ED to receive either EGDT for a total of 6 hours post-randomisation, or standard care.

Patients assigned to receive EGDT will be cared for by the dedicated ARISE study team. The patient will receive treatment as per the study protocol for 6 hours with central blood oxygen levels as the target end-point, then receive standard care.

Patients assigned to receive standard care will continue to be cared for by the hospital team in accordance with current best practice.

Patients in both groups will also receive any additional treatment needed, such as antibiotics or surgery.

This study will involve 1600 patients with severe sepsis admitted to the ED from multiple hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection
* The presence of TWO or MORE of the following SIRS criteria:

  * Core temperature < 36.0 degC or > 38.0 degC
  * Heart rate > 90 beats/minute
  * Respiratory rate > 20 breaths/minute or PaCO2 < 32 mmHg or the requirement for mechanical ventilation for an acute process
  * White blood cell count > 12.0 or < 4.0 x109/L or > 10% immature band forms
* Evidence of either refractory hypotension OR hypoperfusion:

  * Refractory hypotension is confirmed by the presence of a systolic blood pressure (SBP) < 90 mmHg or mean arterial pressure (MAP) < 65 mmHg after a 1000ml intravenous (IV) fluid challenge within 60 minutes (including IV fluids administered pre-hospital)
  * Hypoperfusion is confirmed by the presence of a blood lactate concentration greater than or equal to 4.0 mmol/L
* First dose of IV antimicrobial therapy commenced prior to randomisation

Exclusion Criteria:

* Age < 18 years
* Contra-indication to superior vena cava (SVC) CVC insertion
* Contra-indication to blood products (e.g. Jehovah's Witness)
* Inability to commence delivery of the EGDT protocol within 1 hour of randomisation or complete 6 hours of EGDT
* Haemodynamic instability due to active bleeding
* Pregnancy (confirmed or suspected)
* In-patient transfer from another acute health care facility
* An underlying disease process with a life expectancy of < 90 days
* Death is deemed imminent and inevitable
* A "limitation of therapy" order has been documented restricting implementation of the study protocol or the treating clinician deems aggressive care unsuitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2008-10; Primary Completion 2014-07 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure for the study is death from all causes | 90 days

SECONDARY OUTCOMES:
Death from all causes | 28 days, and at ICU and hospital discharge
Quality of life as measured by the SF-36v2, EQ-5D and the AQoL | 6 and 12 months post-randomisation
Duration of ED, ICU and hospital stay | 28 days and 90 days
The need for, and duration of, artificial organ support | 28 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, Principal Investigator — Austin Hospital, Melbourne Australia; Sandra L Peake, Study Chair — The Queen Elizabeth Hospital
Locations (51):
- Australia (42):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Coffs Harbour Hospital, Coffs Harbour, New South Wales
  - St Vincent's Hospital (Sydney), Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Hornsby Hospital, Hornsby, New South Wales
  - Manly Hospital, Manly, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Port Macquarie Base, Port Macquarie, New South Wales
  - Prince of Wales Hospital (Sydney), Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Sydney Adventist hospital, Sydney, New South Wales
  - Tamworth Hospital, Tamworth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston Brisbane, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Modbury Hospital, Modnury, South Australia
  - Bendigo Hospital, Bendigo, Victoria
  - Blacktown Hospital, Blacktown, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Alfred, Prahan, Victoria
  - Central Gippsland (Sale Hospital), Sale, Victoria
  - Joondalup Health Campus, Joondalup, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Finland (2):
  - Helsinki University Hospital, Helsinki, Finland
  - Tampere University Hospital, Tampere, Finland
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong, Hong Hong
  - Pamela Youde Nethersole Eastern Hospital (HK), Chai Wan, Hong Kong
  - The Queen Elizabeth Hospital (HK), Kowloon, Hong Kong
- St. Vincent's University hospital, Dublin, Ireland
- New Zealand (3):
  - Middlemore Hospital, Otahuhu Auckland, Auckland
  - Christchurch Hospital, Christchurch, New Zealand
  - Auckland City Hospital, Auckland

REFERENCES:
- [Derived] Higgins AM, Peake SL, Rinaldo Bellomo AO, Ao DJC, Delaney A, Howe BD, Nichol AD, Webb SA, Williams PJ, Harris AH; ARISE Investigators and the ANZICS Clinical Trials Group. The cost-effectiveness of early goal-directed therapy: an economic evaluation alongside the ARISE trial. Crit Care Resusc. 2023 Oct 18;23(3):329-336. doi: 10.51893/2021.3.OA10. eCollection 2021 Sep 6. PMID 38046082
- [Derived] Higgins AM, Peake SL, Bellomo R, Cooper DJ, Delaney A, Harris AH, Howe BD, Nichol AD, Webb SA, Williams PJ; Australasian Resuscitation in Sepsis Evaluation (ARISE) Investigators and the ANZICS Clinical Trials Group. Quality of Life and 1-Year Survival in Patients With Early Septic Shock: Long-Term Follow-Up of the Australasian Resuscitation in Sepsis Evaluation Trial. Crit Care Med. 2019 Jun;47(6):765-773. doi: 10.1097/CCM.0000000000003762. PMID 30985391
- [Derived] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Derived] Delaney A, Peake SL, Bellomo R, Cameron P, Holdgate A, Howe B, Higgins A, Presneill J, Webb S; ARISE Investigators. Australasian Resuscitation In Sepsis Evaluation trial statistical analysis plan. Emerg Med Australas. 2013 Oct;25(5):406-15. doi: 10.1111/1742-6723.12116. Epub 2013 Sep 9. PMID 24099368